CLINICAL TRIAL: NCT04951739
Title: To Investigate the Incidence of Reflux in Patients After Per-oral Endoscopic Myotomy in Achalasia Cardia Patients
Status: Completed | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: AIG/IEC-BH&R 13/05.2021-01
Record Dates: First submitted 2021-06-01; First posted 2021-07-07 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Achalasia Cardia; Gastroesophageal Reflux
Keywords: Achalasia cardia; Peroral endoscopic myotomy; Gastroesophageal Reflux; oesophageal pH study; oesophageal acidification; High resolution manometry
MeSH Terms: conditions — Esophageal Achalasia; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Achalasia cardia patients - post peroral endoscopic myotomy: All the patients who will undergo peroral endoscopic myotomy for the treatment of achalasia cardia patients.
  Interventions: Procedure: Peroral endoscopic myotomy

INTERVENTIONS:
Procedure: Peroral endoscopic myotomy — Peroral endoscopic myotomy involves an initial incision on the internal lining of the oesophagus. This permits entry of the endoscope to within the wall of the oesophagus, where the muscle will be exposed. The inner layer of the muscle near the lower oesophagal sphincter will be cut (this is termed myotomy). At the conclusion of the procedure, the oesophagal incision will be closed with standard endoscopic clips.

SUMMARY:
Achalasia is a rare motility disorder of the oesophagus that is characterized by aperistalsis of the oesophagal body and dysrelaxation of the lower oesophagal sphincter (LES). Current treatment is palliative, and the aim of the treatment is to diminish the obstructive function of the esophagogastric junction (EGJ). Due to this approach, the most frequent complication post-treatment is gastroesophageal reflux (GER). However, not every treated patient develops GER symptoms and the mechanism behind the occurrence of GER in treated achalasia are unclear. In this study, we aim to Investigate the incidence of reflux in patients after peroral endoscopic myotomy in patients with achalasia cardia.

DETAILED DESCRIPTION:
1. INTRODUCTION- Achalasia is a rare motility disorder of the oesophagus that is characterized by aperistalsis of the oesophagal body and dysrelaxation of the lower oesophagal sphincter (LES). Current treatment is palliative, and the aim of the treatment is to diminish the obstructive function of the esophagogastric junction (EGJ). Due to this approach, the most frequent complication post-treatment is gastroesophageal reflux (GER). However, not every treated patient develops GER symptoms and the mechanism behind the occurrence of GER in treated achalasia are unclear. In this study, we aim to Investigate the incidence of reflux in patients after peroral endoscopic myotomy in patients with achalasia cardia.
2. STUDY OBJECTIVES

   Our hypothesis is those gastroesophageal reflux symptoms in treated patients with achalasia are dependent on retention and fermentation of food due to a reduced clearance by aperistalsis of the oesophageal body rather than the result of actual acid reflux episodes. We expect a difference in gastroesophageal reflux episodes, LES pressure in the treated patients with achalasia that experience gastroesophageal reflux symptoms compared to the the group that does not encounter gastroesophageal reflux symptoms.
3. STUDY POPULATION This observational study has a prospective design. Two groups of study subjects will be included. Treated patients with achalasia with gastroesophageal reflux symptoms and treated patients with achalasia without gastroesophageal reflux symptoms. On the baseline, clinical data will be collected regarding medical history, family history and medical symptoms related to GER or achalasia.In all the included study subjects, several measurements will be done at AIG hospitals, Hyderabad. The duration of the study is dependent on the rate of inclusion of the study subjects but, it is expected that in 6 months, all study subjects will be included.
4. DESIGN AND DURATION OF THE STUDY- It will be a prospective observational study for 6 months.
5. METHODOLOGY

5a. SUBJECT RECRUITMENT - Treated patients with idiopathic achalasia visiting the outpatient clinic will be asked to participate in the study. Only when a study subject has given informed consent, questionnaires concerning demographic and clinical data will be recorded, and measurements will be performed.

5b. RANDOMIZATION AND BLINDING- NO

5c. STUDY METHODS-

5d.STUDY PROCEDURE-

Baseline clinical data will be collected using different questionnaires. The participant will be subjected to the GERD Questionnaire to be sure that he or she is allocated to the correct study group. For this study, all included study subjects will undergo a few measurements. Upper GI endoscopy under conscious sedation will be done, followed by a timed barium oesophagogram &. High-resolution manometry will be done. The barium oesophagography is performed to gain insight into oesophageal emptying and the width of the oesophagus. After peroral endoscopic myotomy has been done, these measurements, including upper GI endoscopy, 24 hours ambulatory pH and impedance testing, High-resolution oesophageal manometry & Timed barium oesophagogram, will be done at 3 months of follow-up.

5e. Study requirements and timeline

The measurements will be performed after cessation of PPIs, H2-antagonists and medications that can influence intestinal motility for one week. To reduce severe symptoms, patients are allowed to take rescue medication in the form of antacids. Furthermore, one day before the measurements, the patients will be restricted to a liquid diet to minimize the stasis of food in the oesophagus. Study subjects will arrive in the morning at the AIG hospital after an overnight fast, with no intake of fluid after midnight except water. If this is not possible, the medication should, of course, be ingested before the measurements. Before the first measurements, patients must have been fasting for four hours, so also no intake of water. UGI endoscopy followed by High-resolution oesophageal manometry later timed barium esophagogram will be done.

The formal investigation for patients with reflux symptoms after one month will be UGI endoscopy, High-resolution oesophageal manometry and 24-hour ambulatory pH-impedance monitoring. Study subjects go home with the pH-impedance catheter in place and will receive a diary to write down their symptoms. During this measurement, the study subject has to drink and eat at everyday moments. Still, there is no restriction concerning the food intake, except again an overnight fast due to the timed barium oesophagography the next day. The following day patients come back to the hospital where the pH-impedance catheter will be removed, and a timed barium oesophagography will be performed, which is the last measurement.

5f. METHODS OF ASSESSMENT-

A)High-Resolution Manometry (HRM)

A water-perfused high-resolution manometry assembly with 21 water-perfused sensors spaced at 1-cm intervals at the position of the esophagogastric junction will be used.

Each sensor is accurate to within 1mmHg, capable of recording transient pressure changes over 6000 mmHg/s, and zeroed to atmospheric pressure. The high-resolution manometry assembly will be introduced transnasal and positioned to record from hypopharynx to stomach with about five intragastric sensors. Data are analyzed using Solar high-resolution manometry software (Medical Measurement Systems, Enschede, The Netherlands).

B) pH- impedance monitoring

A pH-impedance catheter will be introduced transnasally. A 2.1-mm outer diameter study catheter comprised of six electrode pairs measuring intraluminal impedance at 3, 5, 7, 9, 15 and 17 cm above the LES and an ISFET pH sensor, placed 5 cm above the LES will be used. Before and after recording the pH electrode will be calibrated using standard buffers of pH seven and pH 1. The catheter will be positioned in such a way that the pH sensor is located 5 cm above the LES, which is based on manometry readings.

C) Analysis of the data of the HRM and pH-impedance monitoring

For analysis of the data obtained with HRM and pH-impedance measurement, MMS software (Enschede, The Netherlands) Will be used.The HRM will give insight into the esophageal function. It provides information on the contractile activity of the oesophagal body and the esophagogastric junction, including the LES. Therefore it helps distinguish transient LES relaxation (TLESRs), which occurs in GERD, from pseudo relaxation of the LES by shortening the oesophagal body. pH impedance monitoring provides information on oesophagal bolus transit. GER is characterized by TLESRs and a retrograde moving decrease in impedance with an abrupt drop in pH levels followed by normalization of the impedance and pH. In the case of fermentation, there is a slight and longer decrease in impedance and pH. The pH-impedance monitoring will also record all reflux episodes, both acid as non-acid, during the 24-hours measurement. During the analysis of the data of the pH-impedance monitoring, reflux symptoms will be correlated with acid and non-acid reflux episodes. A positive correlation is declared if a specific reflux symptom is preceded by a reflux episode within two minutes. The analysis will be done manually for all the patients as the risk of false-positive is more with the automated analysis. Oesophageal acidification patterns observed during pH-impedance monitoring.

1. Acid reflux with average clearance: rapid pH drop to below 4, drop rate ≥one pH unit per second, lasting between 10 s and 5 min.
2. Acid reflux with delayed clearance: rapid pH drop to below 4, drop rate≥one pH unit per second, lasting longer than 5 min.
3. Acid fermentation: slow pH drop to below 4, drop rate <1 pH unit per minute, prevailing longer than 5 min most specific for achalasia cardia. Automated analysis can count these refluxes as false positive and can misdiagnose fermentation as reflux after POEM.
4. Stasis of recently ingested acidic food or drink: pH drops to below four during meal/drink, pH below 4 persisting longer than 5 min after meal/drink.
5. Unclassified: pH drop below 4, not meeting criteria for any of the acid patterns described above.

D) Timed barium esophagram

A maximal tolerable amount of low-density barium sulphate must be ingested by the study subjects in 30-45 s without regurgitation or aspiration. After ingestion of low-density barium sulphate, oesophageal stasis will be determined at 1, 2 and 5 minutes with the study subject upright in a slight left posterior position. The distance from the tapered distal oesophagus to the top of the barium column and the maximal diameter of the oesophagus is measured.

E) Questionnaires

* Eckardt score, which is the sum of symptom scores for dysphagia, regurgitation, chest pain, and weight loss. Each symptom is scored from 0 to 3. The minimum score is 0, and the maximum score is 12. Pre and post values will be recorded.
* The validated Achalasia Disease-Specific Quality-of-Life questionnaire (Achalasia- DSQoL). Pre and post POEM values will be recorded.
* The validated Gastroesophageal Reflux Disease Questionnaire (GERDQ) is a self-assessment questionnaire that can be used for the diagnosis and follow-up of gastroesophageal reflux disease. It measures both symptoms and the impact of symptoms on a person's daily life.

  5g. STOPPING OR DISCONTINUATION CRITERIA- NOT APPLICABLE

  6. OUTCOME MEASURES Three-month post peroral endoscopic myotomy

  7. SAMPLE SIZE CALCULATION- Sample size- 50 patients Expected outcomes - 18- 28 per cent is likely to be symptomatic post POEM surgery, and true reflux incidence maybe around 5- 10 per cent. Considering incidence for GERD population from south India, around 8 per cent sample size will be about 50, with the study's power as 80 per cent, with 95 per cent confidence interval and 5 per cent margin of error.

  8. STATISTICAL ANALYSIS- Data will be expressed as median and percentile values (5th, 25th, 75th and 95th percentiles). Depending on the normality of distribution, we will use either paired Student's t-test or Mann-Whitney U test for paired comparison. Likewise, we will use a one-way analysis of variance with Tukey test or Kruskal-Wallis, followed by Dunn's test as appropriate. The upper limit of normal will be defined as the 95th percentile of expected values. For PSPW index and MNBI thresholds, we will use the 5th and 25th percentile values. P≤0.05 will be considered statistically significant.

  9. ETHICAL JUSTIFICATION OF THE STUDY All patients of Achalasia patients who undergo palliative treatment in the form of peroral endoscopic measurement will be tested after the procedure at 3 months. It will give us insight into the true incidence of GERD and also will determine their therapy based on the phenotype they fit in.

ELIGIBILITY:
Inclusion Criteria:

A- Treated achalasia patients with gastroesophageal reflux symptoms

* Diagnosis of idiopathic achalasia confirmed by oesophageal manometry that shows the following criteria:
* Aperistalsis or simultaneous contractions in the oesophageal body.
* Impaired relaxation of the Lower oesophageal sphincter
* Treatment of achalasia with per-oral endoscopic myotomy (POEM)
* The minimum total score on the Gastroesophageal Reflux Disease Questionnaire (GERDQ) of ≥ 8.
* Gastroesophageal symptoms after treatment lasting more than three months.
* Age 18-80 years.
* Written informed consent.

B- Treated achalasia patients without gastroesophageal reflux symptoms

Diagnosis of idiopathic achalasia confirmed by oesophagal manometry that shows the following criteria:

* Aperistalsis or simultaneous contractions in the oesophageal body.
* Impaired relaxation of the Lower oesophageal sphincter
* Treatment of achalasia with per-oral endoscopic myotomy (POEM)
* The maximum total score on the Gastroesophageal Reflux Disease Questionnaire (GERDQ) of < 8.
* Age 18-80 years.
* Written informed consent.

EXCLUSION CRITERIA-

* Pseudoachalasia.
* Upper gastrointestinal malignancy.
* Chagas disease.
* Peptic ulcer disease.
* Inability to stop PPI, H2-receptor antagonist or prokinetic drug for two weeks
* Presence of an extremely dilated oesophagus body >5 cm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Treated achalasia patients with and without gastroesophageal reflux symptoms visiting the outpatient clinic of the Gastroenterology Department.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
To Investigate the incidence of reflux in patients after peroral endoscopic myotomy in achalasia cardia patients. | Three months
  To study the incidence of true reflux in patients with achalasia cardia who have undergone peroral endoscopic myotomy with 24 hour ambulatory pH monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Aniruddha P Singh, MBBS,MD,DM, Principal Investigator — AIG hospitals,India; Mohan Ramchandani, MBBS,MD,DM, Study Director — AIG Hospitals,India; Nageshwar Reddy, MBBS,MD,DM, Study Chair — AIG Hospitals,India; Pradev Inavolu, MBBS, MD, DM, Principal Investigator — AIG Hospitals, India; Hardik Rughwani, MBBS, MD, DM, Principal Investigator — AIG Hospitals, India; Neeraj Singla, MBBS, MD, DM, Principal Investigator — AIG Hospitals, India
Locations (1):
- AIG Hospitals, Hyderabad, Telangana, India

REFERENCES:
- [Result] Boeckxstaens GE. The lower oesophageal sphincter. Neurogastroenterol Motil. 2005 Jun;17 Suppl 1:13-21. doi: 10.1111/j.1365-2982.2005.00661.x. PMID 15836451
- [Result] Campos GM, Vittinghoff E, Rabl C, Takata M, Gadenstatter M, Lin F, Ciovica R. Endoscopic and surgical treatments for achalasia: a systematic review and meta-analysis. Ann Surg. 2009 Jan;249(1):45-57. doi: 10.1097/SLA.0b013e31818e43ab. PMID 19106675
- [Result] Lopushinsky SR, Urbach DR. Pneumatic dilatation and surgical myotomy for achalasia. JAMA. 2006 Nov 8;296(18):2227-33. doi: 10.1001/jama.296.18.2227. PMID 17090769
- [Result] Anderson SH, Yadegarfar G, Arastu MH, Anggiansah R, Anggiansah A. The relationship between gastro-oesophageal reflux symptoms and achalasia. Eur J Gastroenterol Hepatol. 2006 Apr;18(4):369-74. doi: 10.1097/00042737-200604000-00009. PMID 16538107
- [Result] Crookes PF, Corkill S, DeMeester TR. Gastroesophageal reflux in achalasia. When is reflux really reflux? Dig Dis Sci. 1997 Jul;42(7):1354-61. doi: 10.1023/a:1018873501205. PMID 9246028
- [Result] van Herwaarden MA, Samsom M, Smout AJ. Prolonged manometric recordings of oesophagus and lower oesophageal sphincter in achalasia patients. Gut. 2001 Dec;49(6):813-21. doi: 10.1136/gut.49.6.813. PMID 11709516
- [Result] Shoenut JP, Micflikier AB, Yaffe CS, Den Boer B, Teskey JM. Reflux in untreated achalasia patients. J Clin Gastroenterol. 1995 Jan;20(1):6-11. doi: 10.1097/00004836-199501000-00004. PMID 7884182
- [Result] Katzka DA, Sidhu M, Castell DO. Hypertensive lower esophageal sphincter pressures and gastroesophageal reflux: an apparent paradox that is not unusual. Am J Gastroenterol. 1995 Feb;90(2):280-4. PMID 7847301
- [Result] Novais PA, Lemme EM. 24-h pH monitoring patterns and clinical response after achalasia treatment with pneumatic dilation or laparoscopic Heller myotomy. Aliment Pharmacol Ther. 2010 Nov;32(10):1257-65. doi: 10.1111/j.1365-2036.2010.04461.x. Epub 2010 Sep 25. PMID 20955445
- [Result] Shoenut JP, Duerksen D, Yaffe CS. A prospective assessment of gastroesophageal reflux before and after treatment of achalasia patients: pneumatic dilation versus transthoracic limited myotomy. Am J Gastroenterol. 1997 Jul;92(7):1109-12. PMID 9219779
- [Result] Spechler SJ, Souza RF, Rosenberg SJ, Ruben RA, Goyal RK. Heartburn in patients with achalasia. Gut. 1995 Sep;37(3):305-8. doi: 10.1136/gut.37.3.305. PMID 7590421
- [Result] Eckardt VF, Aignherr C, Bernhard G. Predictors of outcome in patients with achalasia treated by pneumatic dilation. Gastroenterology. 1992 Dec;103(6):1732-8. doi: 10.1016/0016-5085(92)91428-7. PMID 1451966
- [Result] Rohof WO, Hirsch DP, Kessing BF, Boeckxstaens GE. Efficacy of treatment for patients with achalasia depends on the distensibility of the esophagogastric junction. Gastroenterology. 2012 Aug;143(2):328-35. doi: 10.1053/j.gastro.2012.04.048. Epub 2012 May 2. PMID 22562023
- [Result] Rohof WO, Lei A, Boeckxstaens GE. Esophageal stasis on a timed barium esophagogram predicts recurrent symptoms in patients with long-standing achalasia. Am J Gastroenterol. 2013 Jan;108(1):49-55. doi: 10.1038/ajg.2012.318. Epub 2012 Sep 25. PMID 23007004
- [Result] Vaezi MF, Baker ME, Achkar E, Richter JE. Timed barium oesophagram: better predictor of long term success after pneumatic dilation in achalasia than symptom assessment. Gut. 2002 Jun;50(6):765-70. doi: 10.1136/gut.50.6.765. PMID 12010876
- [Result] Kwiatek MA, Kahrilas K, Soper NJ, Bulsiewicz WJ, McMahon BP, Gregersen H, Pandolfino JE. Esophagogastric junction distensibility after fundoplication assessed with a novel functional luminal imaging probe. J Gastrointest Surg. 2010 Feb;14(2):268-76. doi: 10.1007/s11605-009-1086-1. PMID 19911238
- [Result] Hemmink GJ, Bredenoord AJ, Weusten BL, Timmer R, Smout AJ. Does acute psychological stress increase perception of oesophageal acid? Neurogastroenterol Motil. 2009 Oct;21(10):1055-e86. doi: 10.1111/j.1365-2982.2009.01327.x. Epub 2009 May 15. PMID 19453516
- [Derived] Singh AP, Singla N, Budhwani E, Januszewicz W, Memon SF, Inavolu P, Nabi Z, Jagtap N, Kalapala R, Lakhtakia S, Darisetty S, Reddy DN, Ramchandani M. Defining "true acid reflux" after peroral endoscopic myotomy for achalasia: a prospective cohort study. Gastrointest Endosc. 2024 Feb;99(2):166-173.e3. doi: 10.1016/j.gie.2023.08.008. Epub 2023 Aug 19. PMID 37598862